CLINICAL TRIAL: NCT03125057
Title: A Pilot Study of Hemoporfin Photodynamic Therapy in Children (7-14 Years Old) With Port-wine Stain
Brief Title: A Pilot Study of Hemoporfin PDT in Children With Port-wine Stain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Fudan-Zhangjiang Bio-Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: HMME-C1610
Record Dates: First submitted 2017-04-19; First posted 2017-04-24 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Port-wine Stain
MeSH Terms: conditions — Port-Wine Stain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- low light dose (Experimental): PDT is applied to the patients at low light dose : power density of 60mW/cm2 for 20 minutes
  Interventions: Drug: Hemoporfin PDT
- high light dose (Experimental): PDT is applied to the patients at high light dose : power density of 75mW/cm2 for 20 minutes
  Interventions: Drug: Hemoporfin PDT

INTERVENTIONS:
Drug: Hemoporfin PDT — Photodynamic therapy is performed using hemoporfin. Hemoporfin（5mg/kg）is infused for 20 minutes, followed by light illumination at 10 minutes from the start of infusion. Different light dose of PDT is applied to the patients.

SUMMARY:
This pilot study aims to evaluate the efficacy and safety of hemoporfin photodynamic therapy (PDT) with different light doses for port-wine stain (PWS） in 7-14 years old children. The population pharmacokinetics of hemoporfin in children will be investigated as well.

ELIGIBILITY:
Inclusion Criteria:

* Children with clinical diagnosis of PWS；
* Age range: 7 to 14 years-old；
* Voluntarily participated and Written informed consent signed

Exclusion Criteria:

* Therapy area located outside of head and neck;
* Other skin diseases that might interfere with the efficacy evaluation;
* Therapy area was previously received isotope or PDT or other treatment which might interfere with the efficacy evaluation;
* Allergy to porphyrins and analogues; Photosensitivity; Porphyria; Allergic constitution;
* Scar diathesis;
* Immunocompromised conditions;
* Electrocardiographic abnormalities or organic heart diseases;
* Coagulation disorders;
* Hepatic or renal functions abnormal (alanine aminotransferase or aspartate transaminase or total bilirubin > 1.5 upper limit of normal [ULN], or serum creatinine or blood urea nitrogen > 1.5 ULN);
* Psychiatric diseases; Severe endocrinopathies;
* Previous therapy of PWS within the last 4 weeks;
* Participation in any clinical studies within the last 4 weeks;
* Be judged not suitable to participate the study by the investigators

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2017-08-02 (Actual); Primary Completion 2020-05-10 (Actual); Study Completion 2020-05-10 (Actual)

PRIMARY OUTCOMES:
Response rate | week 8
  proportion of patients achieving at least some improvement (color blanching from the baseline >= 20%)

CONTACTS AND LOCATIONS:
Overall Officials: Lin Ma, MD, Principal Investigator — Bejing Children's Hospital, Capital Medical University; Jining Tao, Study Director — Shanghai Fudan-Zhangjiang Bio-Pharmaceutical Co., Ltd.
Locations (1):
- Beijing Children's Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No